CLINICAL TRIAL: NCT02113098
Title: Effects of Treadmill Gait Training With Adding Load on Lower Limb of Individuals With Stroke
Brief Title: Effects of Treadmill Gait Training With Loading in Individuals With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Ana Raquel Rodrigues Lindquist, PhD, PhD, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 488.293
Record Dates: First submitted 2014-04-10; First posted 2014-04-14 (Estimated); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Stroke; Gait Disorders, Neurologic
Keywords: Stroke; Gait; Rehabilitation
MeSH Terms: conditions — Stroke; Gait Disorders, Neurologic | interventions — Exercise Test

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treadmill, ankle load (Experimental): The experimental group will perform gait training on a treadmill with added load to the non-paretic lower limb
  Interventions: Other: Treadmill, ankle load
- Treadmill (Active Comparator): The control group (active comparator) will perform gait training on a treadmill
  Interventions: Other: Treadmill

INTERVENTIONS:
Other: Treadmill, ankle load — The experimental group will perform gait training on a treadmill (Gait Trainer 2®) with added load to the ankle of the non-paretic lower limb, plus physical therapy correction for restore gait symmetry. The intervention will last 30 minutes, in nine sessions for two weeks
  Arms: Treadmill, ankle load
Other: Treadmill — The control group (active comparator) will perform gait training on a treadmill (Gait Trainer 2®) with physical therapy correction for restore gait symmetry. The intervention will last 30 minutes, in nine sessions for two weeks
  Arms: Treadmill

SUMMARY:
The purpose of this study is to determine whether the add load on non-paretic lower limb of individuals that suffer a stroke, while walking on a treadmill, is effective for restore gait symmetry of these individuals, in a subacute phase of stroke.

DETAILED DESCRIPTION:
This is a randomized and blinded clinical trial, in which participants are being randomly divided into experimental group and control group, in order to verify the effects of adding load on gait symmetry after stroke. 40 individuals will participate, and the calculation of sample size was performed from the ratio variable symmetry of swing time, based on previous study. Whereas about 15% of individuals could give up to participate in the study during their course (dropout rate), we determined a number of 20 participants in each group.

ELIGIBILITY:
Inclusion Criteria:

* First episode of stroke (ischemic or hemorrhagic) which determined unilateral hemiparesis
* Time of lesion less one year
* Able to walk independently by 10 feet on flat surface without the use of assistive devices
* Gait speed less than 0.8 m / s
* Ability to understand and obey simple commands

Exclusion Criteria:

* Instability of cardiac conditions
* Adverse clinical conditions affecting balance and / or gait
* Pain and / or severe discomfort that impede the realization of the proposed activities
* Decompensation in systemic blood pressure, with the systolic and diastolic values above 200 mmHg and 110 mmHg, respectively, before and / or after training
* Submaximal heart rate above the allowed values during training

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Ground reaction force, in Newtons | Until one year after stroke
  Vertical component of ground reaction force, measured using a force platform
Angular displacements of hip, knee and ankle (in degrees) | Until one year after stroke
  Angular gait variables, measured by a system of movement analysis.
Symmetry ratio (swing time of paretic limb/swing time of non-paretic limb) | Until one year after stroke
  Spatiotemporal gait variable, measured by a system of movement analysis

SECONDARY OUTCOMES:
speed (meters/second) | Until one year after stroke
  Spatiotemporal gait variable, measured by a system of movement analysis
double support time (in seconds) | Until one year after stroke
  Spatiotemporal gait variable, measured by a system of movement analysis
step length (in meters) | Until one year after stroke
  Spatiotemporal gait variable, measured by a system of movement analysis
stride length (in meters) | Until one year after stroke
  Spatiotemporal gait variable, measured by a system of movement analysis

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana S Ribeiro, MSc, Principal Investigator — Universidade Federal do Rio Grande do Norte
Locations (1):
- Universidade Federal do Rio Grande do Norte, Natal, Rio Grande do Norte, Brazil

REFERENCES:
- [Derived] E Silva EMGS, Ribeiro TS, da Silva TCC, Costa MFP, Cavalcanti FADC, Lindquist ARR. Effects of constraint-induced movement therapy for lower limbs on measurements of functional mobility and postural balance in subjects with stroke: a randomized controlled trial. Top Stroke Rehabil. 2017 Dec;24(8):555-561. doi: 10.1080/10749357.2017.1366011. Epub 2017 Aug 31. PMID 28859603